CLINICAL TRIAL: NCT05305404
Title: Dexamethasone to Target Stress and Immune System Changes During Early Abstinence in Individuals With Alcohol Use Disorder (AUD)
Brief Title: Dexamethasone to Target Stress and Immune System Mechanisms Underlying Alcohol Craving
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Helen Fox, PhD, Assistant Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AA029735 (NIH)
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Alcohol Use Disorder
Keywords: Stress; Dexamethasone; Immune system; Cortisol
MeSH Terms: conditions — Alcoholism | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: This is a two arm assignment where participants are randomized to a single dose dexamethasone (1.5mg) or placebo
Who Masked: Participant, Investigator
Masking Description: Study is double blind, where participants and investigators are blind to the medication assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guanfacine (Active Comparator): single dose of dexamethasone (1.5mg) administered orally
  Interventions: Drug: Dexamethasone Oral
- Placebo (Placebo Comparator): single dose of placebo administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone Oral — 1.5mg oral dexamethasone to be administered once at 11:00PM
  Other Names: Decadron, Dexamethasone Intensol, Dexasone, Solurex, and Baycadron.
  Arms: Guanfacine
Drug: Placebo — oral placebo to be administered once at 11:00PM
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled, proof of concept laboratory study to recruit N=70 (35 Males / 35 Females) non-treatment seeking, heavy drinkers with alcohol use disorder (AUD). It is hypothesized that randomization to 1.5mgs dexamethasone versus placebo will decrease alcohol craving during stress by decreasing basal cortisol, increasing anti-inflammatory cytokine levels and potentially normalizing the immune response to stress.

ELIGIBILITY:
Inclusion Criteria:

* Non-treatment seeking heavy drinking men and women with AUD
* Age range 18-55,
* Body Mass Index (BMI) of 18-35
* Positive ethylglucuronide (EtG) urine toxicology screen for alcohol
* Able to provide informed written and verbal consent
* Able to read English and complete study evaluations
* Good health as verified by screening examination.

Exclusion Criteria:

* Meet criteria for Substance Use Disorder (SUD) or other psychoactive substances, excluding nicotine
* Unable to remain abstinent for five days
* Need for a medically assisted detoxification
* Regular use of steroids, anticonvulsants, sedatives/hypnotics, prescription analgesics, other anti-hypertensives, anti-arrythmics, antiretroviral medications, tricyclic antidepressants, naltrexone, disulfiram, and any other psychoactive medications with the exception of stabilization on Selective Serotonin Re-uptake Inhibitors (SSRIs)
* Psychotic or severely psychiatrically disabled
* Significant underlying medical conditions which would be of potential harm
* Pregnancy or breast feeding women;
* Women using monophasic contraceptives
* Electrocardiogram (EKG) evidence of clinically significant conduction abnormalities, (Bazlett's corrected QT (QTc) interval of >450 msec for men and QTc>470 msec for women).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-06-23 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Alcohol craving as assessed using subjective report following stress exposure | Change from baseline to +5 minutes following stress exposure
  The 8-item Alcohol Urges Questionnaire (AUQ) will be used to measure alcohol craving. There are 8 items, each with a Likert scale response from 1 to 7 (1: Strongly Disagree, 7: Strongly Agree). Total possible score of 56. The higher the score the higher the alcohol craving
Alcohol craving as assessed using subjective report following stress exposure | Change from baseline to +15 minutes following stress exposure
  The 8-item Alcohol Urges Questionnaire (AUQ) will be used to measure alcohol craving. There are 8 items, each with a Likert scale response from 1 to 7 (1: Strongly Disagree, 7: Strongly Agree). Total possible score of 56. The higher the score the higher the alcohol craving
Alcohol craving as assessed using subjective report following stress exposure | Change from baseline to +30 minutes following stress exposure
  The 8-item Alcohol Urges Questionnaire (AUQ) will be used to measure alcohol craving. There are 8 items, each with a Likert scale response from 1 to 7 (1: Strongly Disagree, 7: Strongly Agree). Total possible score of 56. The higher the score the higher the alcohol craving
Alcohol craving as assessed using subjective report following stress exposure | Change from baseline to +5 minutes following stress exposure
  A visual analog scale will be used to measure alcohol craving. Participants will be required to rate "how much they are craving alcohol right at this moment". The scale will be anchored from 1 to 10 (1: Not at all, 10: Extremely)
Alcohol craving as assessed using subjective report following stress exposure | Change from baseline to +15 minutes following stress exposure
  A visual analog scale will be used to measure alcohol craving. Participants will be required to rate "how much they are craving alcohol right at this moment". The scale will be anchored from 1 to 10 (1: Not at all, 10: Extremely)
Alcohol craving as assessed using subjective report following stress exposure | Change from baseline to +30 minutes following stress exposure
  A visual analog scale will be used to measure alcohol craving. Participants will be required to rate "how much they are craving alcohol right at this moment". The scale will be anchored from 1 to 10 (1: Not at all, 10: Extremely)
Hypothalamic-Pituitary-Adrenal (HPA)-axis response to stress exposure as assessed by cortisol | Change from baseline to +5 minutes following stress exposure
  4mls of plasma cortisol will be collected following exposure to stress
HPA axis response to stress exposure as assessed by cortisol | Change from baseline to +15 minutes following stress exposure
  4mls of plasma cortisol will be collected following exposure to stress
HPA axis response to stress exposure as assessed by cortisol | Change from baseline to +30 minutes following stress exposure
  4mls of plasma cortisol will be collected following exposure to stress
HPA axis response to stress exposure as assessed by Adrenocorticotropic Hormone (ACTH) | Change from baseline to +5 minutes following stress exposure
  4mls of plasma ACTH will be collected following exposure to stress
HPA axis response to stress exposure as assessed by ACTH | Change from baseline to +15 minutes following stress exposure
  4mls of plasma ACTH will be collected following exposure to stress
HPA axis response to stress exposure as assessed by ACTH | Change from baseline to +30 minutes following stress exposure
  4mls of plasma ACTH will be collected following exposure to stress
Immune system response to stress exposure as assessed by peripheral cytokines | Change from baseline to +5 minutes following stress exposure
  4mls of plasma Interleukin (IL)-10 will be collected following exposure to stress
Immune system response to stress exposure as assessed by peripheral cytokines | Change from baseline to +15 minutes following stress exposure
  4mls of plasma IL-10 will be collected following exposure to stress
Immune system response to stress exposure as assessed by peripheral cytokines | Change from baseline to +30 minutes following stress exposure
  4mls of plasma IL-10 will be collected following exposure to stress
Immune system response to stress exposure as assessed by peripheral cytokines | Change from baseline to +5 minutes following stress exposure
  4mls of plasma Interleukin 1 receptor antagonist (IL1-ra) will be collected following exposure to stress
Immune system response to stress exposure as assessed by peripheral cytokines | Change from baseline to +15 minutes following stress exposure
  4mls of plasma IL1-ra will be collected following exposure to stress
Immune system response to stress exposure as assessed by peripheral cytokines | Change from baseline to +30 minutes following stress exposure
  4mls of plasma IL1-ra will be collected following exposure to stress
Immune system response to stress exposure as assessed by peripheral cytokines | Change from baseline to +5 minutes following stress exposure
  4mls of plasma IL-6 will be collected following exposure to stress
Immune system response to stress exposure as assessed by peripheral cytokines | Change from baseline to +15 minutes following stress exposure
  4mls of plasma IL-6 will be collected following exposure to stress
Immune system response to stress exposure as assessed by peripheral cytokines | Change from baseline to +30 minutes following stress exposure
  4mls of plasma IL-6 will be collected following exposure to stress
Immune system response to stress exposure as assessed by peripheral cytokines | Change from baseline to +5 minutes following stress exposure
  4mls of plasma Tumor Necrosis Factor alpha (TNFa) will be collected following exposure to stress
Immune system response to stress exposure as assessed by peripheral cytokines | Change from baseline to +15 minutes following stress exposure
  4mls of plasma TNFa will be collected following exposure to stress
Immune system response to stress exposure as assessed by peripheral cytokines | Change from baseline to +30 minutes following stress exposure
  4mls of plasma TNFa will be collected following exposure to stress
Immune system response to stress exposure as assessed by peripheral cytokines | Change from baseline to +5 minutes following stress exposure
  4mls of plasma Tumor Necrosis Factor Receptor 1 (TNFR1) will be collected following exposure to stress
Immune system response to stress exposure as assessed by peripheral cytokines | Change from baseline to +15 minutes following stress exposure
  4mls of plasma TNFR1 will be collected following exposure to stress
Immune system response to stress exposure as assessed by peripheral cytokines | Change from baseline to +30 minutes following stress exposure
  4mls of plasma TNFR1 will be collected following exposure to stress

SECONDARY OUTCOMES:
Anxiety as assessed using subjective report following stress exposure | Change from baseline to +5 minutes following stress exposure
  A visual analog scale will be used to measure anxiety. Participants will be required to rate "how nervous, anxious or jittery they are feeling at this moment". The scale will be anchored from 1 to 10 (1: Not at all, 10: Extremely)
Anxiety as assessed using subjective report following stress exposure | Change from baseline to +15 minutes following stress exposure
  A visual analog scale will be used to measure anxiety. Participants will be required to rate "how nervous, anxious or jittery they are feeling at this moment". The scale will be anchored from 1 to 10 (1: Not at all, 10: Extremely)
Anxiety as assessed using subjective report following stress exposure | Change from baseline to +30 minutes following stress exposure
  A visual analog scale will be used to measure anxiety. Participants will be required to rate "how nervous, anxious or jittery they are feeling at this moment". The scale will be anchored from 1 to 10 (1: Not at all, 10: Extremely)
Negative Mood as assessed using subjective report following stress exposure | Change from baseline to +5 minutes following stress exposure
  The Differential Emotion Scale will be used to measure negative mood. Participants will be required to rate on a 5-point scale the extent to which an emotional word describes the way they feel at the current time. 1: not at all, 5: Extremely
Negative Mood as assessed using subjective report following stress exposure | Change from baseline to +15 minutes following stress exposure
  The Differential Emotion Scale will be used to measure negative mood. Participants will be required to rate on a 5-point scale the extent to which an emotional word describes the way they feel at the current time. 1: not at all, 5: Extremely
Negative Mood as assessed using subjective report following stress exposure | Change from baseline to +30 minutes following stress exposure
  The Differential Emotion Scale will be used to measure negative mood. Participants will be required to rate on a 5-point scale the extent to which an emotional word describes the way they feel at the current time. 1: not at all, 5: Extremely

CONTACTS AND LOCATIONS:
Overall Officials: Helen C Fox, PhD, Principal Investigator — Stony Brook Renaissance School of Medicine
Locations (1):
- The Health Sciences Center, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No